CLINICAL TRIAL: NCT03752242
Title: An Exploratory Trial to Evaluate the Clinical Effectiveness of a Topical Application of BMX-010 in Subjects With Acne Vulgaris.
Brief Title: Evaluation of Topical Application of BMX-010 in Subjects With Acne Vulgaris.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment stopped for chemistry work on investigational product.
Sponsor: BioMimetix JV, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMX-DERM-203
Record Dates: First submitted 2018-11-15; First posted 2018-11-23 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Masking Description: In Part A, all subjects will receive study drug and this is Open Label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMX-010 0.03% (Experimental): Approximately 30 subjects will receive BMX-010 0.03% for 7-28 days to be applied topically to Acne of the face.
  Interventions: Drug: BMX-010 0.3%

INTERVENTIONS:
Drug: BMX-010 0.3% — Safety and efficacy of BMX-010 in topical treatment of acne.

SUMMARY:
This is an exploratory Phase 2 trial of BMX-010 in patients with Acne Vulgaris which will be conducted in two parts.

DETAILED DESCRIPTION:
Part A is designed to confirm the optimal formulation, strength, and dosing frequency of the study drug in patients with Acne. Up to 60 subjects will be enrolled in this part.

Part B is designed to be a randomized, double-blind trial studying the optimal formulation, strength, and dosing frequency of BMX-010 as determined in Part A, compared to Placebo in patients with Acne. Up to 150 subjects will be enrolled in this part. In both parts, adult subjects with Acne will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age;
2. A clinical diagnosis of mild to severe facial Acne Vulgaris; Subjects may also have acne at other body sites;
3. Screening and Baseline IGA score > 2 (greater than or equal to 2);
4. Willing to refrain from using any topical or systemic treatments for inflammatory skin disease, other than the investigational product;
5. Candidate for topical treatment of Acne;
6. If a cleanser, moisturizer or sunscreen is needed during the study, Subjects must be willing to use only allowed cleansers, moisturizers, sunscreens, or moisturizer/sunscreen combination products. If the subject wears makeup they must agree to use non-comedogenic makeup.
7. Females of child-bearing potential must have a negative urine pregnancy test within 48 hours prior to the first drug administration;
8. Females of child-bearing potential must be willing to use 2 methods of contraception deemed adequate by the investigator (for example, oral contraceptive pills plus a barrier method) through the trial and for 1 month thereafter to be eligible for, and continue participation in, the study;
9. Ability to complete the study in compliance with the protocol, including agreement in writing to apply study product only to the assigned areas; and
10. Ability to understand and provide written informed consent.

Exclusion Criteria:

1. Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive;
2. Use of androgen receptor blockers (such as spironolactone or flutamide);
3. Severe cystic acne, acne conglobate, acne fulminans, or secondary acne;
4. Use of phototherapy devices, energy-based devices, adhesive cleansing strips, or cosmetic procedures (e.g., facials, peeling, comedo extraction) in the past week;
5. Presence of beard or excessive facial hair at Screening which would interfere with the study treatments or study assessments and refusal to remove for duration of study;
6. Prior or current concomitant therapies that would interfere with assessments in the study;
7. Subjects with any underlying disease that the Investigator deems uncontrolled, and poses a concern for the subject's safety while participating in the study;
8. Use of anti-inflammatory medications, salicylic acid; corticosteroids, antibiotics, antibacterials (including benzoyl peroxide-containing products [e.g., benzamycin]), retinoids; other topical acne treatments (e.g., photodynamic therapy, medicated soaps such as those containing benzoyl peroxide, salicylic acid, sulfur, or sodium sulfacetamide) in the past 2 weeks;
9. Oral retinoid use (e.g., isotretinoin) within 6 months prior to baseline or vitamin A supplements greater than 10,000 units/day within 6 months of baseline;
10. Concomitant skin disease that could confound clinical evaluations or increase risk to the subject;
11. Use of medicated make-up (including anti-aging make-up) throughout the study;
12. Use during the study of 1) systemic steroids, 2) topical retinoids to the face, 3) antibiotics known to impact acne, 4) immunosuppressive agents, or immunomodulators;
13. Facial use of 1) topical steroids, 2) topical anti-inflammatory agents, 3) topical antimycotics, 4) any topical acne treatments or 4) topical antibiotics;
14. Use of medicated cleansers on the face (throughout the study);
15. Use of topical astringents or abrasives, medical topical preparations (prescription and OTC products) within 2 days prior to Baseline and throughout the study;
16. Systemic or skin infection requiring antimicrobial therapy;
17. Systemic chemotherapy or radiotherapy within 4 weeks of the Baseline Visit;
18. Immunocompromise of any cause, known human immunodeficiency virus infection, or acquired immunodeficiency syndrome;
19. Pregnancy, planned pregnancy, lactation, or inadequate contraception as judged by the investigator;
20. Active drug or alcohol dependence;
21. Significant acute or chronic medical, neurological, or psychiatric illness that, in the judgment of the investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study;
22. Previous clinical trial participation for the indication being treated in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado Skin Care, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BMX-010 0.03%
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BMX-010 0.03%
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2
Inflammatory Lesions [Mean (Standard Deviation); unit: count] | 12 (8)
Non-Inflammatory Lesions [Mean (Standard Deviation); unit: count] | 26 (24)

OUTCOME MEASURES:

1. Primary Outcome: Determine Whether the Optimum Frequency of Topical Application of BMX-010 0.03% is Once a Day or Twice a Day Day or Twice Per Day for a Treatment Interval of 7 to 28 Days.
Description: Assessed by change in the 5-point Investigator Global Assessment (IGA), compared amongst the group that is treated once a day versus twice a day. This will be measured weekly from Days 1-28. The Investigator global assessment scale is a global assessment of disease as the time of evaluation. The lowest number on the scale (0) is clear from disease while the highest number (4) is severe disease. Scores on the scale are: 0, 1, 2, 3, 4
Time Frame: 28 days
Population: 2 subjects enrolled and both were treated twice a day, so we were unable to determine this outcome. We will report the IGA scores collected, however this data is insufficient to determine optimal dosing (once a day or twice a day), since the only subjects enrolled were treated twice a day.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BMX-010 0.03%
Number analyzed (Participants) | 2
score on a scale | 2.5 (.5)

2. Primary Outcome: Evaluate the Efficacy of BMX-010 in Treatment of Acne Vulgaris.
Description: Assessed by change in the 5-point Investigator Global Assessment (IGA). This will be measured weekly from Days 1-28, followed by a final assessment two weeks after dosing ends at day 43. Assessed by change in the 5-point Investigator Global Assessment (IGA), compared amongst the group that is treated with study drug versus with placebo. This will be measured weekly from Days 1-28. The Investigator global assessment scale is a global assessment of disease as the time of evaluation. The lowest number on the scale (0) is clear from disease while the highest number (4) is severe disease. Scores on the scale are: 0, 1, 2, 3, 4
Time Frame: 43 days
Population: all of the subjects enrolled in the study
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BMX-010 0.03%: Subjects will receive BMX-010 0.03% to be applied topically to Acne of the face for up to 28 days
  BMX-010 0.3%: Safety and efficacy of BMX-010 in topical treatment of acne.
Arm/Group | BMX-010 0.03%
Number analyzed (Participants) | 2
score on a scale | 2.5 (.5)

3. Secondary Outcome: Assess the Mean Percent Reduction Change in Inflammatory Lesion Counts From Baseline to End of Study.
Description: Inflammatory lesions will be counted at each study visit and the total change in the count of lesions will be assessed from baseline to day 43.
Time Frame: 43 days
Population: Total number of subjects enrolled (n=2)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | BMX-010 0.03%
Number analyzed (Participants) | 2
percentage of change | 7.5 (5.5)

4. Secondary Outcome: Assess the Mean Percent Reduction Change in Noninflammatory Lesion Counts From Baseline to End of Study.
Description: Non-Inflammatory lesions will be counted at each study visit.
Time Frame: 43 days
Population: the total number of subjects enrolled (n=2)
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- BMX-010 0.03%: Subjects will receive BMX-010 0.03% be applied topically to Acne of the face for up to 28 days.
  BMX-010 0.3%: Safety and efficacy of BMX-010 in topical treatment of acne.
Arm/Group | BMX-010 0.03%
Number analyzed (Participants) | 2
percentage of change | 25 (25)

ADVERSE EVENTS:
Time Frame: Treatment Period through Day 43 Final Clinic Visit
Arm/Group | BMX-010 0.03%
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
The clinical trial was stopped after enrollment of 2 subjects for re-formulation of investigational product. Therefore, due to the small sample size data is uninterpretable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT03752242/Prot_000.pdf